CLINICAL TRIAL: NCT00357747
Title: A Phase I Study of AEG35156 in Combination With Docetaxel in Patients With Solid Tumors
Brief Title: AEG35156 and Docetaxel in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I166; CAN-NCIC-IND166 (Other: PDQ); CDR0000481440 (Other: PDQ)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — AEG 35156; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AEG35156 plus docetaxel (Experimental)
  Interventions: Drug: AEG35156; Drug: docetaxel

INTERVENTIONS:
Drug: AEG35156 — After a recommended phase II dose (RPTD) of AEG35156 has been determined with docetaxel 75 mg/m2, patients will be accrued to the RPTD-1 plus docetaxel 100 mg/m2, and possibly RPTD plus docetaxel 100 mg/m2, to determine the RPTD of AEG35156 in combination with docetaxel 100 mg/m2 given every three weeks.
Drug: docetaxel — After a recommended phase II dose (RPTD) of AEG35156 has been determined with docetaxel 75 mg/m2, patients will be accrued to the RPTD-1 plus docetaxel 100 mg/m2, and possibly RPTD plus docetaxel 100 mg/m2, to determine the RPTD of AEG35156 in combination with docetaxel 100 mg/m2 given every three weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. AEG35156 may help docetaxel work better by making tumor cells more sensitive to the drug.

PURPOSE: This phase I trial is studying the side effects and best dose of AEG35156 when given together with docetaxel in treating patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and define the recommended phase II dose of AEG35156 in combination with docetaxel in patients with solid tumors.

Secondary

* Determine the qualitative and quantitative toxicities of AEG35156 and docetaxel and define duration and reversibility of those toxicities.
* Determine the pharmacokinetic profile of this regimen.
* Assess, preliminarily, the antitumor activity of this regimen in patients with measurable disease.
* Assess the pharmacodynamic effects of AEG35156 administration on X-linked inhibitor of apoptosis protein (XIAP) levels and apoptosis in peripheral blood mononuclear cells and, in selected patients, in tumor tissue.
* Evaluate M30/M65 cytokeratin 18 level, a marker of apoptosis/necrosis of epithelial tumors, in these patients.

OUTLINE: This is a multicenter, open-label, dose-escalation study of AEG35156.

Patients receive AEG35156 IV continuously on days -2 and -1. Patients then receive AEG35156 IV continuously over 24 hours on days 1, 8, and 15. Beginning with course 2, patients also receive docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AEG35156 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Blood is collected at baseline and periodically during study treatment for pharmacokinetic and pharmacodynamic assessment.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Locally advanced, metastatic, or recurrent disease that is refractory to standard curative therapy or for which no curative therapy exists
* Clinically and/or radiographically documented disease
* Docetaxel single-agent therapy must be a reasonable treatment option
* No newly diagnosed CNS metastases

  * Previously treated, intracranial disease that has been stable for ≥ 6 months allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* Creatinine normal
* AST and ALT ≤ 1.5 times upper limit of normal
* PT or INR normal
* PTT normal
* No known bleeding disorder
* No preexisting peripheral neuropathy ≥ grade 2
* No prior serious allergic reaction to taxanes (e.g., paclitaxel or docetaxel)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious illness or medical condition that would be aggravated by treatment or preclude study requirements, including any of the following:

  * Serious uncontrolled infection
  * Significant cardiac dysfunction
  * Significant neurological disorder

PRIOR CONCURRENT THERAPY:

* No more than 2 prior chemotherapy regimens for metastatic or recurrent disease
* No more than 1 prior adjuvant chemotherapy regimen
* No more than 1 prior taxane-containing regimen
* At least 4 weeks since prior chemotherapy and recovered
* At least 4 weeks since prior external-beam radiotherapy provided < 30% of marrow-bearing areas are irradiated*
* At least 4 weeks since prior investigational agents or new anticancer therapy
* At least 2 weeks since prior hormonal therapy or immunotherapy
* At least 2 weeks since prior surgery and recovered
* No prior nephrectomy
* No concurrent anticoagulant therapy in therapeutic doses

  * Nontherapeutic dose anticoagulant therapy (e.g., 1 mg warfarin once daily) allowed
* No other concurrent experimental drugs or anticancer therapy
* No other concurrent cytotoxic therapy or radiotherapy

  * Small-volume, nonmyelosuppressive palliative radiotherapy allowed NOTE: *Exceptions are made for prior low-dose non-myelosuppressive radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-06-09 (Actual); Primary Completion 2006-09-26 (Actual); Study Completion 2010-06-07 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity evaluated according to the NCI CTCAE version 3.0 | Every 3 weeks
Response and progression using RECIST criteria | Every 6 weeks
Response duration measured from the time complete response or partial response (whichever is first recorded) is documented until the first date that recurrent or progressive disease is objectively documented | Every 3 months
  After completion of protocol therapy, patients with PR/CR ongoing assessed q3 months until relapse.
Stable disease duration measured from the time of start of therapy until the criteria for progression are met | Every 3 months
  After completion of protocol therapy, patients with ongoing SD assess q 3months until progression.
Pharmacokinetics | cycle 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, MD, Study Chair — Jewish General Hospital
Locations (3):
- Canada (3):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No